CLINICAL TRIAL: NCT03092622
Title: Effects of Aerobic Interval Training on Cardiac Function, With Special Focus on Pulmonary Pressures and Right Sided Function, in Patients With Chronic Obstructive Pulmonary Disease and Hypoxemia
Brief Title: Aerobic Interval Training in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Hypoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013/2129
Record Dates: First submitted 2017-02-22; First posted 2017-03-28 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary; Hypoxia
Keywords: Exercise Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary; Hypoxia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise training (Experimental): Outpatients treadmill interval training, 4x4 minutes with 3 minutes in between at lower intensity. 3 sessions weekly for 10 weeks to a total of 30 sessions.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise training intervention as described earlier.

SUMMARY:
Patients with severe Chronic Obstructive Pulmonary Disease (COPD) and low oxygen levels in the blood are at risk of developing pulmonary hypertension and strain on the right side of the heart, both of which are known to increase symptoms and worsen prognosis It is not fully established whether interval exercise training in patients with severe COPD and concomitant low oxygen levels is beneficial.

This study aims to evaluate the effects of aerobic interval exercise training in patients with severe COPD and low oxygen levels in the blood, with a particular emphasis on such effects on the cardiovascular system and pulmonary circulation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD)
* Forced Expiratory Volume 1 second (FEV1) <60% of predicted
* FEV1%FVC <70 % of predicted (FVC = Forced Vital Capacity)
* Qualify for Long term oxygen therapy (LTOT), or presence of significant desaturation on exercise.

Exclusion Criteria:

* Unstable ischaemic heart disease or valvular heart disease.
* Active malignant disease.
* Substance abuse.
* Physical or mental disability that prevents participation in the exercise programme or testing.
* Pregnancy.
* Exacerbation of COPD or respiratory tract infection last 6 weeks before.
* Completed pulmonary rehabilitation programme or other organised exercise programme last 3 month
* Use of high doses of systemic steroids.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary artery pressure | Change from baseline at 10 weeks
  Examined by right heart catheterisation

OTHER OUTCOMES:
Cardiac function | Change from baseline at 10 weeks
  assessed by echocardiography
Cardiac function | Change from baseline at 10 weeks
  assessed by right heart catheterisation
Respiratory function | Change from baseline at 10 weeks
  assessed by spirometry
Respiratory function | Change from baseline at 10 weeks
  assessed by diffusion capacity,
Respiratory function | Change from baseline at 10 weeks
  assessed by arterial blood gas
Functional capacity | Change from baseline at 10 weeks
  assessed by shuttle walk test
Functional capacity | Change from baseline at 10 weeks
  assessed by 6 minute walk test
Symptoms | Change from baseline at 10 weeks
  COPD Assessment Test (CAT)
Quality of life | Change from baseline at 10 weeks
  St George Respiratory Questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Toril A Nagelhus Hernes, phd prof, Study Chair — Norwegian University of Science and Technology; Sigurd Steinshamn, md prof, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Lungemedisinsk Avdeling & Hjertemedisinsk Avdeling, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No